CLINICAL TRIAL: NCT01811667
Title: Clinical Study on Efficacy and Safety of the mTor Rapamycin Inhibitor Found in the Complex Vascular Malformations
Brief Title: Efficacy and Safety of the Mammalian Target of Rapamycin (mTor Rapamycin) Inhibitor in Vascular Malformations
Acronym: vasca-LM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: vasca-LM
Record Dates: First submitted 2012-10-05; First posted 2013-03-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Cardiovascular Abnormalities
Keywords: Vascular Abnormalities
MeSH Terms: conditions — Cardiovascular Abnormalities | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sirolimus (Experimental): Seric level between 10 to 15 ng/ml Pills for the adults and liquid for the children. Twice a day.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus
  Other Names: rapamycin

SUMMARY:
The phosphatidylinositol 3-kinase (PI3Kinase)/Protein Kinase B (AKT)/mammalian target of rapamycin (mTor) pathway plays a role on the development and the lymphatic-vascular organisations.

The investigators want to study the efficacy and the safety of Rapamycin, an mTor inhibitor.

DETAILED DESCRIPTION:
The complex vascular malformations induce chronical pains and organic dysfunctions causing significant morbidity and mortality. Therefore, the investigators need to establish guidelines in order to treat these pathologies. Standard treatments such as surgery or interventional radiology are of limited efficacy and related to a high level of recurrences as well as complications. Recent preclinical studies have shown the important role of the PI3Kinase/AKT/mTor pathway on the development and the lymphatic-vascular organisations suggesting an appealing therapeutic target to treat patients with complex vascular malformations.

The aim of this clinical study is to prospectively evaluate the efficacy and the safety of the Rapamycin, an mTOR inhibitor, to treat children and adults with microcystic lymphatic malformations, general lymphatics abnormalities (GLA) or complex vascular malformations for which conventional therapies as surgery or sclerotherapy are ineffective or associated with high risk of important complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complex vascular abnormalities to be threat by a systemic therapy
* Patients must have adequate liver function (LDL-cholesterol, triglycerides,…)
* Patients must have adequate organ function: neutrophils >1500/mm³, Hb > 8,0 g et platelets> 50.000/mm³ (no platelets limits for the Kasabach Merritt syndrome)
* Patients must have adequate renal function(normal creatinin depending on the age), clearance > 70 ml/min/1.73m² and Urin Protein Creatinine ratio <0.3 g.
* Karnofsky or Landry > 50

Exclusion Criteria:

* Dental equipments or prosthesis interfering onto a radiological examen
* Other uncontrolled medical condition (uncontrolled diabetes, hypertension…)
* Concomitant drugs such as inhibitors/inducers of cytochrome P450 3A4 (CYP3A4)
* Immunocompromised patients, including known seropositivity for HIV
* Digestive problems modifying the absorption of Rapamycin (gastric tube feeding accepted)
* Pregnant or nursing (lactating) women
* Prior treatment with phosphatidylinositol 3-kinase (PI3K) and/or mTOR inhibitors

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Time of duration of the treatment.(Efficacy) | up to 12 months

SECONDARY OUTCOMES:
The number of adverse events observed | up to 12 months
  With Common Toxicity Criteria for Adverse Effects version 3

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Boon, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Brussels Capital, Belgium